CLINICAL TRIAL: NCT01630213
Title: Vitamin D and Omega-3 Trial: Ancillary Study (VITAL-Echo) on the Impact of Vitamin D Supplementation on Cardiac Structure and Function
Brief Title: Impact of Vitamin D Supplementation on Cardiac Structure and Function
Acronym: VITAL-Echo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ravi Thadhani, Chief, Division of Nephrology; Director of Clinical Research in Nephrology, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009P-001217
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Disease
Keywords: Vitamin D3; Left ventricular mass; Echocardiography; Left ventricular systolic and diastolic function
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Cholecalciferol; Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 + fish oil/placebo (Active Comparator): Vitamin D3 2000 IU/day and fish oil (840 omega 3-fatty acids; Omacor)(or fish oil placebo)/day
  Interventions: Dietary Supplement: Vitamin D3 + fish oil/fish oil placebo
- Vitamin D3 placebo + fish oil/placebo (Placebo Comparator): Vitamin D3 placebo + fish oil (840 mg of omega 3-fatty acids; Omacor)/fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 placebo + fish oil/fish oil placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 + fish oil/fish oil placebo — Vitamin D3 2000 IU/day and fish oil (840 mg of omega 3-fatty acids; Omacor)/fish oil placebo per day
  Other Names: Cholecalciferol; Omacor
  Arms: Vitamin D3 + fish oil/placebo
Dietary Supplement: Vitamin D3 placebo + fish oil/fish oil placebo — Vitamin D3 placebo/day + fish oil (840 mg of omega 3-fatty acids; Omacor)/fish oil placebo/day
  Other Names: Vitamin D3 placebo; Omacor
  Arms: Vitamin D3 placebo + fish oil/placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is a randomized clinical trial in 20,000 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or fish oil (1 gram of omega-3 fatty acids) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study (VITAL-Echo) is being conducted among participants in VITAL and will examine whether vitamin D compared to placebo: (1) reduces left ventricular (LV) mass in elderly individuals as measured with 2-dimensional echocardiography and (2) improves LV systolic and diastolic function as measured with tissue Doppler echocardiography.

DETAILED DESCRIPTION:
Recognition of the biological effects of vitamin D on cardiovascular function has been growing. The main objective of the parent trial (VITAL) is to evaluate the effects of vitamin D on cardiac events but is focused on atherothrombotic events and does not specifically address vitamin D effects on LV mass. In ambulatory individuals, LV mass is a key cardiac structural feature and increases in LV mass are frequently accompanied by diastolic dysfunction. This study leverages the existing infrastructure of the parent VITAL trial to perform cardiac imaging studies on a subset of subjects who will be randomized to vitamin D3 (n=500) or placebo (n=500). Echocardiography is a noninvasive, widely accessible tool to evaluate cardiac structure and function. Cardiac echo imaging visits will take place at baseline (pre-randomization), and then after 2 years, at the Massachusetts General Hospital (MGH). The acronym VITAL-Echo reflects the link to the parent VITAL trial and an ancillary investigation of vitamin D versus placebo on LV mass and function as measured by echocardiography. The effect of fish oil supplementation on these parameters will be evaluated as a secondary endpoint, thereby taking advantage of the factorial design of the parent trial.

ELIGIBILITY:
Participants in VITAL (NCT 01169259) who meet the following criteria are eligible to participate in this ancillary study:

Inclusion:

* Willingness to participate in ancillary study of VITAL to undergo cardiac echocardiography (baseline and at 3 years) and sign informed consent to participate in the ancillary study
* Live in the greater Boston area (within 60 miles of MGH)

Exclusion:

* Have a pacemaker, prosthetic valve(s), surgical wires or other devices that could alter the echocardiographic image findings.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1025 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular (LV) mass | Baseline and 2 years
  Primary aim is to examine whether vitamin D supplementation reduces LV mass in elderly individuals, using 2-dimensional echocardiography.

SECONDARY OUTCOMES:
Change in LV systolic/diastolic function | Baseline and 2 years
  LV systolic and diastolic function using tissue Doppler echocardiography (2 D Echo will be used to measure ejection fraction in systole; E wave, E' E deceleration time, pulmonary vein inflow patterns in diastole; tissue doppler will measure S' in systole and E' in diastole; Speckle tracking will measure global longitudinal strain, LV torsion in systole and oeak LV untwisting rate in diastole).
Change in LV mass | Baseline and 2 years
  To examine whether vitamin D supplementation with/without fish oil supplementation reduces LV mass in elderly individuals, using 2-dimensional echocardiography.
Change in LV systolic/diastolic function | Baseline and 2 years
  Effect of Vitamin D with/without fish-oil on LV systolic and diastolic function using tissue Doppler echocardiography (as above).

CONTACTS AND LOCATIONS:
Overall Officials: Ravi I Thadhani, MD, MPH, Principal Investigator — Massachusetts General Hospital; Thomas J Wang, MD, Principal Investigator — Vanderbilt University Medical Center; Michael H Picard, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chandra A, Picard MH, Huang S, Gupta DK, Agusala K, Buring JE, Lee IM, Cook NR, Manson JE, Thadhani RI, Wang TJ. Impact of Vitamin D3 Versus Placebo on Cardiac Structure and Function: A Randomized Clinical Trial. J Am Heart Assoc. 2022 Nov;11(21):e025008. doi: 10.1161/JAHA.121.025008. Epub 2022 Oct 26. PMID 36285795